CLINICAL TRIAL: NCT03342625
Title: High Intensity Focused Ultrasound Treatment of Breast Tumors. BRIFU Study (Breast Resection By HIFU)
Brief Title: High Intensity Focused Ultrasound Treatment of Breast Tumors. BRIFU Study
Acronym: BRIFU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB 2015-01; ID-RCB number : 2017-A01490-53 (Other: ANSM)
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Female
Keywords: High intensity focused ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Focused Ultrasound (Experimental): High Intensity Focused Ultrasound for the treatment of breast tumors, guided by MRI
  Interventions: Device: High Instensity Focused Ultrasound

INTERVENTIONS:
Device: High Instensity Focused Ultrasound — High Intensity Focused Ultrasound guided by MRI
  Other Names: HIFU

SUMMARY:
Monocentric prospective study evaluating the efficacy of High intensity focused ultrasound (HIFU) in breast tumors.

DETAILED DESCRIPTION:
Incidence of breast cancer increases with the lifetime of the population, and represents an important socio-economic issue. Diagnosis and treatment are major public health issues. High Instensity Focused Ultrasound (HIFU) is a minimally invasive technique which decreases the risk of post-treatment complications and allows shorter hospitalization times. This technology is also remarkable for the absence of limitation related to the dose delivered, which makes it possible to repeat if necessary and the absence of ionizing radiation both for the treatment itself and for its guidance (MRI).

The main objective is to evaluate the efficacy of HIFU for the treatment of breast tumors, based on histological criteria.

Indication :

Histologically invasive ductal carcinoma, T0, with unifocal or plurifocal lesion, with or without associated microcalcifications, measuring 15 mm maximum on ultrasound and clinical N0.

Course of the study :

* Signature of consent,
* Clinical and radiological assessment at Baseline,
* Realization of the HIFU procedure under local anesthesia and sedation (J0),
* Total or partial mastectomy depending on the lesion (between D2 and D8),
* Consultation with surgeon (J30),

Number of patients :

15 patients will be included in this pilot study. If no success is observed, the study will be stopped and the technique considered inefficient. If there are one or more successes, an Independant Data Monitoring Committee (IDMC) will meet to propose an additional trial if necessary with the data from this trial.

ELIGIBILITY:
Inclusion Criteria :

1. Histologically proven infiltrating ductal carcinoma with the analysis of hormone receptors, tumor grade, Her-2 expression.
2. T0 lesion, unifocal or plurifocal, with or without micro-calcifications associated, measuring 15 mm maximum major axis on ultrasound.
3. Clinical N0.
4. Bra cup size greater than or equal to B.
5. Markable and identifiable lesion in MRI.
6. Indication of partial or total mastectomy in case of multifocal lesions or extensive calcification associated with axillary surgery.
7. Breast assessment performed by a referent radiologist: Mammography, ultrasound, clinical examination.
8. No contraindication to MRI.

Exclusion Criteria :

1. Infiltrating lobular carcinoma and Pure ductal carcinoma in situ.
2. Bilateral lesion.
3. Non-detectable MRI lesions, within 10 mm of the skin, greater than 15 mm on ultrasound.
4. Unifocal palpable tumor.
5. Cup size bra equal to A.
6. Cutaneous lesion on the breast to be treated by HIFU.
7. Impossibility of ventral decubitus immobility, extended arm, during 1 hour.
8. Pregnant or postpartum patient.
9. Patient participating in another interventional clinical trial within 30 days of enrollment and during the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of HIFU for the treatment of breast tumors, based on histological criteria | Day 30
  * Complete success: absence of viable invasive tumor cells on histological analysis.
  * Incomplete success: Partial tumor destruction of the invasive contingent, unhealthy margins due to underestimation of tumor volume before treatment or imperfect targeting of focused ultrasound. Incomplete successes will be considered as failures. The persistence of an in situ quota alone will be considered as success.
  * Failure: presence of viable invasive tumor cells in the treated area.

SECONDARY OUTCOMES:
Feasibility of non-invasive pre-surgical identification of the tumor area to be resected (palpation by the surgeon of the focused ultrasound ablation zone) | Day 2, 8
Immediate complications of focused ultrasound | Day 30
Pain (visual analogue scale) experienced by patients during the sedation procedure, until surgery. | Day 0, 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean PALUSSIERE, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided